CLINICAL TRIAL: NCT00897052
Title: Survival Prediction in HNSCC Based on Gene Expression Profiles From FFPE Tissues
Brief Title: Gene Expression Profiles in Predicting Survival of Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0511; VU-VICC-HN-0511; VU-VICC-IRB-040509
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — To identify gene expression profile associated with survival from formalin-fixed paraffin embedded tissue samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: microarray analysis — Assay RNA obtained from archived formalin fixed paraffin embedded tissue samples
Other: laboratory biomarker analysis — The gene expression data will be linked to the clinical information in order to generate profile of recurrence and survival as a biomarker.

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict survival of patients with head and neck cancer.

PURPOSE: This laboratory study is assessing gene expression profiles in predicting survival of patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify gene expression profiles associated with survival by DNA microarray assay analysis using RNA from formalin-fixed paraffin-embedded tissue samples from patients with squamous cell carcinoma of the head and neck treated on clinical trial RTOG-9501.

OUTLINE: Formalin-fixed paraffin-embedded tissue samples are analyzed by DNA microarray analysis for gene expression profiling.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell carcinoma of the head and neck, including 1 of the following sites:

  * Hypopharynx
  * Larynx
  * Oral cavity
  * Oropharynx
* Stage II-IV disease
* Must have received treatment on clinical trial RTOG-9501
* Formalin-fixed paraffin-embedded tissue samples available

Exclusion Criteria:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prior patients who participated on clinical trial RTOG-9501
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Identification of gene expression profiles used to predict survival as assessed by DNA microarray analysis | at time of surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center